CLINICAL TRIAL: NCT02002845
Title: A Retrospective Multicenter Investigation of the Use of the da Vinci® Surgical System in Non-Tumor Based TORS Procedures
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: Non-Tumor based TORS procedure
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Subjects Who Have Undergone Benign Non-tumor TORS Procedures Using the da Vinci Surgical System
Keywords: Tongue base resection, partial glossectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Robotic arm: Patient who have undergone benign non-tumor TORS procedures using the da Vinci Surgical System
  Interventions: Device: robotic surgery using the da Vinci Surgical System

INTERVENTIONS:
Device: robotic surgery using the da Vinci Surgical System

SUMMARY:
A retrospective multicenter investigation of the use of the da Vinci® Surgical System in Non-Tumor Based TORS Procedures. The study objectives are to evaluate the safety and effectiveness of the da Vinci Surgical System in subjects undergoing Benign Non-tumor procedures.

DETAILED DESCRIPTION:
Primary Effectiveness Endpoint:

• Ability to complete procedure without a need for conversion to a non-robotic approach

Safety Endpoint:

Assessment of adverse events through post-operative follow-up including but not limited to:

• Bleeding

▪ Mortality

Additional endpoints evaluated may include:

* Procedure times
* Length of hospital stay
* Volume of tissue resected
* Use of tissue sealants

ELIGIBILITY:
Inclusion Criteria:

* The specific surgical procedure involved a lingual tonsillectomy, tongue base resection, or a partial glossectomy procedure.
* Subject was ≥18 years of age at the time of procedure

Exclusion Criteria:

* Subject underwent a benign non-tumor TORS procedure that did not involve either a lingual tonsillectomy, tongue base resection or partial glossectomy.
* Subject underwent a TORS procedure for oropharyngeal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone benign non-tumor TORS procedures using the da Vinci Surgical System
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | intra-operative
  Ability to complete procedure without a need for conversion to a non-robotic approach
Primary Safety endpoint | up to 30 days after surgery
  Assessment of adverse events through post-operative follow-up including but not limited to:
  • Bleeding
  ▪ Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Mehendale, MS, Study Director — Intutive Surgical
Locations (3):
- United States (3):
  - Middlesex Hospital, Middletown, Connecticut
  - St. Jose Mercey Health System, Ypsilanti, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania